CLINICAL TRIAL: NCT04289103
Title: A Phase 3, Multicenter, Open Label, Study to Evaluate the EFficacy and SaFEty of Leukotac® (Inolimomab) in Pediatric Patients With Steroid Resistant Acute Graft Versus Host Disease (SR-aGvHD)
Brief Title: Evaluation of EFficacy and SaFEty of Leukotac (Inolimomab) in Pediatric Patients With SR-aGvHD
Acronym: EiFFEL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ElsaLys Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INO-108
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Steroid Refractory GVHD
MeSH Terms: interventions — inolimomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inolimomab/Leukotac (Experimental): * Patient screening phase - Patients diagnosed with aGvHD will be identified. Only patients with SR-aGvHD will be finally included in the study.
  * Treatment phase - Leukotac will be given up to D28
  * Primary Follow-up phase - Patient's response (CR and PR) will be evaluated at D29 post inclusion. Patients will then be followed for survival, long-term safety and chronic GvHD occurrence during 6 months after inclusion
  Interventions: Biological: Inolimomab (Leukotac)

INTERVENTIONS:
Biological: Inolimomab (Leukotac) — * Patient screening phase - Patients diagnosed with aGvHD will be identified. Only patients with SR-aGvHD will be finally included in the study.
  * Treatment phase - Leukotac will be given up to D28
  * Primary Follow-up phase - Patient's response (CR and PR) will be evaluated at D29 post inclusion. Patients will then be followed for survival, long-term safety and chronic GvHD occurrence during 6 months after inclusion.

SUMMARY:
A Phase 3, Multicenter, open label, study to Evaluate the EFficacy and SaFEty of Leukotac® (inolimomab) in pediatric patients with steroid resistant acute Graft versus Host Disease (SR-aGvHD)

ELIGIBILITY:
Inclusion Criteria:

* Patients who develop a first episode of aGvHD stage ≥ II (Przepiorka et al., 1995), resistant to a first line therapy with steroids (lack of improvement after 5 days or progression after 3 days of treatment with corticosteroids at 2 mg/Kg methylprednisolone equivalent dose)
* Age 28 days to < 18 years old
* Allo-HSCT with any type of donor, stem cell source, GVHD prophylaxis or conditioning regimen
* Patients receiving Allo-HSCT for any indication (i.e. malignant or non-malignant disease)
* Signature of informed and written consent by the patient and/or by the patient's legally acceptable representative(s)

Exclusion Criteria:

* Isolated stage 1 skin SR-aGvHD
* Overlap chronic GvHD as defined by the NIH Consensus Criteria (Jagasia MH, 2015)
* Acute GvHD after donor lymphocytes infusion (DLI)
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal
* Other systemic drugs than corticosteroids for GvHD treatment (including extra-corporeal photopheresis). Drugs already being used for GvHD prevention (e.g. calcineurin inhibitors) are allowed.
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy
* Known allergy or intolerance to Leukotac of one of its ingredients
* Pregnancy: positive urinary or blood test in female of childbearing potential; lactation; absence of effective contraceptive method for female and male of childbearing potential
* Other ongoing interventional protocol that might interfere with

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Overall response | Day 29 post inclusion
  Complete response + very good partial response + partial response

IPD SHARING:
Plan to Share IPD: No